CLINICAL TRIAL: NCT07200895
Title: Investigation of the Acute Effects of Inspiratory Muscle Training at Different Intensities on Vital Signs and Peripheral and Respiratory Muscle Strength in Male Smokers
Brief Title: Acute IMT Intensity Effects in Male Smokers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FATMA DİLARA AKAR ÇAMYAR (Other)
Responsible Party: Sponsor-Investigator, FATMA DİLARA AKAR ÇAMYAR, Principal Investigator, Biruni University
Organization: Biruni University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BiruniU-IMT2025
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Smokers
Keywords: Inspiratory muscle training; breathing exercise; respiratory muscle strength; smoking
MeSH Terms: conditions — Smoking | interventions — Maximal Respiratory Pressures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30% MIP IMT (Experimental): Single supervised session of inspiratory muscle training at 30% of maximal inspiratory pressure (MIP) using a threshold device; 3 sets × 30 breaths (~15 minutes) following a standardized diaphragmatic-breathing warm-up.
  Interventions: Device: Inspiratory Muscle Training (30% MIP)
- 60% MIP IMT (Experimental): Single supervised session of inspiratory muscle training at 60% of maximal inspiratory pressure (MIP) using a threshold device; 3 sets × 30 breaths (~15 minutes) following the same standardized warm-up.
  Interventions: Device: Inspiratory Muscle Training (60% MIP)

INTERVENTIONS:
Device: Inspiratory Muscle Training (30% MIP) — Single supervised session of threshold-loaded inspiratory muscle training set at 30% of baseline maximal inspiratory pressure (MIP); 3 sets × 30 breaths (~15 minutes) following a standardized diaphragmatic-breathing warm-up.
  Arms: 30% MIP IMT
Device: Inspiratory Muscle Training (60% MIP) — Single supervised session of threshold-loaded inspiratory muscle training set at 60% of baseline maximal inspiratory pressure (MIP); 3 sets × 30 breaths (~15 minutes) following the same standardized warm-up.
  Arms: 60% MIP IMT

SUMMARY:
Acute IMT Intensity Effects in Male Smokers

DETAILED DESCRIPTION:
Cigarette smoking can impair respiratory muscle function by reducing inspiratory strength and endurance; Inspiratory Muscle Training (IMT) is a rehabilitative strategy that uses resistive breathing to strengthen the diaphragm and accessory inspiratory muscles. It may temporarily influence autonomic responses and muscle performance. This randomised, parallel-group study will investigate the immediate effects of two IMT intensities in male smokers. Thirty-four male participants who currently smoke will be randomly assigned to one of two groups: IMT at 30% of maximal inspiratory pressure (MIP) or IMT at 60% of MIP. Prior to IMT, all participants will complete a standardised diaphragmatic breathing warm-up (3 sets of 10 repetitions; approximately 5 minutes). IMT will be administered with a threshold device (e. g., Powerbreathe®), with each group performing 3 sets of 30 breaths at the assigned intensity over approximately 15 minutes under supervision. Participants will be monitored for transient discomfort or fatigue. Outcomes will be assessed immediately before and after the session. These will include respiratory muscle strength (MIP, maximal expiratory pressure, MEP), peripheral muscle performance (handgrip strength in both dominant and non-dominant hands), and vital signs (heart rate, oxygen saturation, respiratory rate, systolic and diastolic blood pressure), along with perceived exertion using the Borg scale. The primary outcome will be a change in MIP (cmH₂O and % predicted); secondary outcomes will include changes in MEP, handgrip strength, vital signs, and perceived exertion. Data will be analysed using appropriate paired and independent tests (parametric or non-parametric based on distributional checks) in IBM SPSS v 27. By comparing low- and higher-intensity IMT within a single supervised session, the study aims to identify a practical early-intervention intensity that can acutely enhance inspiratory muscle function in male smokers and potentially inform broader pulmonary rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Male, 18-25 years of age.
* Current cigarette smoker for ≥1 year (regular use).
* No known acute or chronic medical condition.

Exclusion Criteria:

* History of any musculoskeletal injury that may limit participation.
* History of chest pain during physical activity.
* Current use of any medication.
* Symptoms of dizziness or balance loss.
* Diagnosis of hemophilia or history of vascular/cardiovascular disease affecting circulation.
* Presence of any acute illness at screening or on the test day.
* Inability to complete the procedures due to physical limitation.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in Maximal Inspiratory Pressure (MIP), cmH₂O and % predicted | Baseline (pre-session) to immediately post-session (within ~5 minutes after IMT)
  MIP will be measured using a calibrated mouth pressure meter/threshold device per standard procedures with a nose clip and from residual volume. The primary endpoint is the within-participant change (post-pre) expressed in cmH₂O and as % predicted based on reference equations. Higher values indicate greater inspiratory muscle strength.

SECONDARY OUTCOMES:
Change in Maximal Expiratory Pressure (MEP), cmH₂O and % predicted | Baseline to immediately post-session
  MEP will be assessed with the same device from total lung capacity. Endpoint is post-pre change (cmH₂O and % predicted). Higher values indicate greater expiratory muscle strength.
Change in Handgrip Strength (dominant and non-dominant), kg | Baseline to immediately post-session
  Assessed with a calibrated hand dynamometer (e.g., Jamar). Best of three trials for each hand recorded. Endpoint is post-pre change (kg).
Change in Heart Rate, Change in Respiratory Rate, Change in Oxygen Saturation, Change in Systolic and Diastolic Blood Pressure, Change in Perceived Exertion | Baseline to immediately post-session
  * Measured at rest using a pulse oximeter or cardiac monitor after 3-5 minutes seated rest. Endpoint is post-pre change (bpm).
  * Counted over 60 seconds at rest. Endpoint is post-pre change (breaths/min).
  * Measured by pulse oximetry with the participant seated and at rest. Endpoint is post-pre change (%).
  * Automated sphygmomanometer, seated, appropriate cuff size, two readings averaged if needed. Endpoint is post-pre change (mmHg).
  * Global rating of exertion collected at rest (pre) and within 1-2 minutes after IMT. Endpoint is post-pre change (points).

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The team is evaluating repository options and consent language for de-identified IPD sharing.

REFERENCES:
- [Background] Tanriverdi A, Kahraman BO, Ozsoy I, Ozpelit E, Savci S. Acute effects of inspiratory muscle training at different intensities in healthy young people. Ir J Med Sci. 2021 May;190(2):577-585. doi: 10.1007/s11845-020-02353-w. Epub 2020 Aug 26. PMID 32851483
- [Background] Rodrigues F, Araujo AA, Mostarda CT, Ferreira J, de Barros Silva MC, Nascimento AM, Lira FS, De Angelis K, Irigoyen MC, Rodrigues B. Autonomic changes in young smokers: acute effects of inspiratory exercise. Clin Auton Res. 2013 Aug;23(4):201-7. doi: 10.1007/s10286-013-0202-1. Epub 2013 Jun 28. PMID 23812534